CLINICAL TRIAL: NCT00238407
Title: Docetaxel and Cisplatin Chemotherapy Followed by Radiochemotherapy in Patients With Inoperable, Locally Advanced Esophageal Cancer, A Multicenter Phase II Trial
Brief Title: Docetaxel, Cisplatin, and Radiation Therapy in Treating Patients With Locally Advanced Esophageal Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 76/02; EU-20529
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Active Comparator): Patients receive docetaxel IV over 30-60 minutes and cisplatin IV over 1 hour on days 1, 22, 43, 50, 57, 64, and 71. Beginning on day 43 (week 7) of chemotherapy, patients undergo radiotherapy once daily, 5 days a week, for 7 weeks.
  Interventions: Drug: Docetaxel and Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Docetaxel and Cisplatin — Patients receive docetaxel IV over 30-60 minutes and cisplatin IV over 1 hour on days 1, 22, 43, 50, 57, 64, and 71.
Radiation: Radiotherapy — Beginning on day 43 (week 7) of chemotherapy, patients undergo radiotherapy once daily, 5 days a week, for 7 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Docetaxel and cisplatin may also make tumor cells more sensitive to radiation therapy. Giving docetaxel and cisplatin together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel and cisplatin together with radiation therapy works in treating patients with locally advanced esophageal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the local tumor-control rate in patients with locally advanced, unresectable esophageal cancer treated with docetaxel, cisplatin, and radiotherapy.

Secondary

* Determine the feasibility of this regimen in these patients.
* Determine the adverse reactions of this regimen in these patients.
* Determine local- and distant-failure and time to local- and distant-failure in patients treated with this regimen.
* Determine overall survival of patients treated with this regimen.
* Determine the long-term survival rate in patients treated with this regimen.
* Determine whether early improvement of dysphagia is a predictive marker in patients treated with this regimen.
* Determine quality of life and clinical benefit in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 30-60 minutes and cisplatin IV over 1 hour on days 1, 22, 43, 50, 57, 64, and 71. Beginning on day 43 (week 7) of chemotherapy, patients undergo radiotherapy once daily, 5 days a week, for 7 weeks.

Quality of life is assessed at baseline, at day 22 and 43 during treatment, and then every 3 months for 1 year after completion of study treatment.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal cancer, including the gastroesophageal junction

  * Squamous cell or adenocarcinoma
  * Unresectable disease
* Meets 1 of the following staging criteria by endoscopic ultrasound:

  * Cervical (supraclavicular) lesion, meeting 1 of the following stages:

    * TX, N+ disease
    * T3-4, NX disease
    * TX, NX, M1a* disease
  * Thoracic (celiac) lesion, meeting 1 of the following stages:

    * Unresectable T4, NX disease
    * TX, NX, M1a* disease
  * Locally advanced resectable tumors, inoperable due to medical reasons NOTE: *M1a requires unequivocal abnormality on staging CT scan/endosonography
* No T1-2, N0 disease
* All tumors encompassable in 1 radiation field
* No tumor with esophagotracheal fistula

PATIENT CHARACTERISTICS:

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine clearance > 60 mL/min

Cardiovascular

* No myocardial infarction within the past 3 months
* No New York Heart Association class III or IV congestive heart failure
* No unstable angina pectoris
* No significant arrhythmias
* No other severe cardiovascular disease

Immunologic

* No uncontrolled active infection
* No active autoimmune disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No definite contraindication to corticosteroids
* No uncontrolled diabetes mellitus
* No pre-existing peripheral neuropathy > grade 1
* No significant neurologic or psychiatric disorder, including psychotic disorders, dementia, or seizures, that would preclude giving informed consent
* No other serious underlying medical condition that would preclude study participation
* No other prior or concurrent malignancy except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Radiotherapy

* No prior radiotherapy to the chest

Other

* More than 30 days since prior experimental treatment in another clinical trial
* No other concurrent experimental drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-03; Primary Completion 2008-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without local failure measured 6 months after completion of study treatment | 6 months

SECONDARY OUTCOMES:
Adverse reactions measured after completion of study treatment | 6 months
Successful completion of therapy measured after completion of study treatment | 6 months
Dysphagia as measured 6 months after completion of study treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Razvan Popescu, MD, Study Chair — Hirslanden Klinik Aarau; Thomas Ruhstaller, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (10):
- Switzerland (10):
  - Hirslanden Klinik Aarau, Aarau
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital, Liestal
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - City Hospital Triemli, Zurich

REFERENCES:
- [Result] Ruhstaller T, Templeton A, Ribi K, Schuller JC, Borner M, Thierstein S, von Moos R, Pederiva S, Lohri A, Lombriser N, von Briel C, Koeberle D, Popescu R. Intense therapy in patients with locally advanced esophageal cancer beyond hope for surgical cure: a prospective, multicenter phase II trial of the Swiss Group for Clinical Cancer Research (SAKK 76/02). Onkologie. 2010;33(5):222-8. doi: 10.1159/000305094. Epub 2010 Apr 9. PMID 20502056